CLINICAL TRIAL: NCT00840957
Title: Pharmaco Kinetic and Pharmacokinetic-Pharmacodynamic Variability of Infliximab
Brief Title: Pharmaco Kinetic Variability of Infliximab in Rheumatoid Arthritis
Acronym: FAKIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: PHRI07-DM / FAKIR; 2007-002752-42 (EudraCT Number); 2007-R21 (Other: CPP); A70582-40 (Other: AFSSAPS)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Rhumatoid arthritis patient currently receiving infliximab
  Interventions: Biological: infliximab

INTERVENTIONS:
Biological: infliximab — chimeric monoclonal antibody to Tumor Necrosis Factor-alpha

SUMMARY:
Infliximab is a chimeric monoclonal antibody directed towards Tumor Necrosis Factor -alpha that is largely used in inflammatory diseases such as rheumatoid arthritis (RA).

A relationship between dose and clinical outcomes was shown in populations of RA patients but there is an interindividual variability of this relationship. At an individual level, this dose-effet relationship can be separated into the dose-concentration (pharmacokinetic or PK) and the concentration-effet (pharmacokinetic-pharmacodynamic or PK-PD) relationships.

Serum trough concentrations of infliximab have been shown to be variable between patients receiving the same treatment regimen. This PK variability may be explained by several factors (e.g. genetic and immunological factors). The concentration-effect relationship may also be variable and the sources of this variability need to be studied as well. To date no detailed infliximab PK analysis has been published. The sources of variability of the dose-effect relationship need to be characterized to optimize infliximab dosing regimen in patients.

The FAKIR study is a multicenter prospective observational study that will focus on patients treated with infliximab. Its aims are:

1. to characterize the PK and PK-PD variability of infliximab in RA, using clinical criteria and biomarkers, assessed over time ;
2. to study the influence of the polymorphism of FCGRT (the gene encoding FcRn) on the PK variability of infliximab; to study the influence of the polymorphism of FCGR3A (the gene encoding Fc gamma RIIIa) on the PK-PD variability of infliximab; and to study the influence of antibodies toward infliximab on the PK and PK-PD variabilities of infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis according to ACR criteria
* Patient already receiving infliximab for more than 14 weeks
* No modification of the dose regimen of infliximab since the last infusion
* No modification of disease modifying anti rheumatic drugs since the last 4 weeks

Exclusion Criteria:

* Surgery scheduled during the duration of the study
* Pregnancy
* infection, malignancy, immune reaction to infliximab or demyelinating diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Characterizing the PK and PK-PD variability of infliximab in RA | 6 to 12 weeks

SECONDARY OUTCOMES:
Studying the relation between FCGRT polymorphism and the PK variability of infliximab; the relation between FCGR3A polymorphism and the PK-PD variability of infliximab; and the relation between ATI and the PK and PK-PD variabilities of infliximab | 6 to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Denis MULLEMAN, MD, Principal Investigator — CHRU de Tours
Locations (6):
- France (6):
  - CHRU de Brest, Brest
  - CHRU de Nantes, Nantes
  - CHR d'Orléans, Orléans
  - CHRU de Poitiers, Poitiers
  - CHRU de Rennes, Rennes
  - CHRU de Tours, Tours

REFERENCES:
- [Result] Ternant D, Ducourau E, Perdriger A, Corondan A, Le Goff B, Devauchelle-Pensec V, Solau-Gervais E, Watier H, Goupille P, Paintaud G, Mulleman D. Relationship between inflammation and infliximab pharmacokinetics in rheumatoid arthritis. Br J Clin Pharmacol. 2014 Jul;78(1):118-28. doi: 10.1111/bcp.12313. PMID 24354889